CLINICAL TRIAL: NCT02124980
Title: Automated Recovery Line for Medication Assisted Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: APT Foundation, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1208010744; R01DA034678 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Drug Dependence; Substance Use Disorders
Keywords: Opioid Substitution Treatment; Cognitive Behavioral Therapy; Mobile Health
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recovery Line plus Treatment-as-Usual (RL+TAU) (Experimental): The Recovery Line is an automated computer-based IVR system that provides CBT-based modules. The RL+TAU condition will include the customized therapeutic recommendations developed in Phase 1, and the contact reminders messages and time frame that maximized system use in Phase 2. Patients will receive an orientation, 24-hour access, encouragement to use the system from clinic staff reminder, and technical assistance line for system problems. Patients will receive 12 weeks of system access.
  Interventions: Behavioral: Recovery Line
- Treatment-as-Usual (No Intervention): Treatment-as Usual involves daily methadone and associated psychosocial services. Patients are required to attend 1 group session per month and are encouraged to attend open drop-in groups available daily covering a range of topics.

INTERVENTIONS:
Behavioral: Recovery Line
  Other Names: Therapeutic interactive voice response; Therapeutic IVR; TIVR
  Arms: Recovery Line plus Treatment-as-Usual (RL+TAU)

SUMMARY:
If shown to be effective, the Recovery Line would provide an inexpensive, transportable, and easy to use treatment to improve substance abuse outcomes for medication assisted treatment. Given the high costs of relapse and continued drug use, improvement of treatment outcomes would provide substantial health, economic, and societal benefits.

DETAILED DESCRIPTION:
Dependence on heroin and prescription pain relievers has almost tripled since 2000, resulting in dramatic increases in opioid dependence treatment admissions. However, among agonist-maintained patients continued drug use is common and associated with high rates of relapse and treatment drop-out. Although counseling has been shown to be effective, it is costly and some patients dislike counseling, others have responsibilities that make attendance difficult, and patients in rural settings often have limited access to psychotherapy. Thus, there is a clear need to develop additional acceptable and cost-effective treatments. Interactive Voice Response (IVR) systems, which have been shown to effectively augment brief interventions for substance abuse, are automated, computer-based systems delivered via phone and use voice or keys to access different menus. IVR systems can be accessed from any phone rather than only specified technology (e.g., smartphones), and offer advantages of low cost, consistent delivery, expanded access, and 24-hour availability of immediate therapeutic intervention. The Recovery Line is a Cognitive Behavioral Therapy (CBT)-based IVR system to reduce substance use in patients receiving opioid agonist maintenance. We recently completed a pilot randomized 4-week trial which showed significant reduction in cocaine use and increased coping skill efficacy, but patients called less time than expected, suggesting methods to improve patient use may further improve efficacy. This Stage Ib application proposes three phases to develop system functions to increase patient system use and to test those functions. The initial two phases will develop customized recommendations and reminders to be used in Phase 3 pilot clinical trial. The Phase 3 trial is a 12-week pilot randomized (N=60), clinical trial with a 3 month post-treatment follow-up to obtain data regarding the feasibility, acceptability and efficacy of the developed Recovery Line (compared to TAU). Efficacy will be evaluated for the two primary outcome domains of the proportion of urine screens negative for illicit drugs and monthly days of illicit drug abstinence. Secondary outcome measures will be retention in treatment and coping skills efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. are at least 18 years old
2. currently receiving methadone maintenance treatment
3. illicit drug use in the past 14 days or a positive urine screen for any tested illicit drug.

Exclusion Criteria:

1. Current suicide or homicide risk
2. meet criteria for Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV current psychotic disorder, or bipolar disorder
3. Unable to read or understand English
4. Unable to complete the study because of anticipated incarceration or move
5. Life-threatening or unstable medical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
urine screens | 6 months
  bi-weekly urine screens negative for illicit drugs
self reported drug use | 6 months
  monthly days of self reported illicit drug abstinence

SECONDARY OUTCOMES:
treatment retention | 6 months
  days retained in methadone treatment
coping behaviors | 6 months
  coping behaviors as measured by the Effectiveness of Coping Behavior Inventory and the Drug Risk Response Test

OTHER OUTCOMES:
patient satisfaction | 6 months
  a semi-structured interview will be used to assess overall satisfaction with methadone services and satisfaction ratings of specific components of treatment
type and amount of health and psychosocial services | 6 months
  the Treatment Services Review is a semistructured used to collect detailed information on receipt of health and psychosocial services outside of the study

CONTACTS AND LOCATIONS:
Locations (1):
- MRU, APT Foundation, Inc, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Moore BA, Buono FD, Printz DMB, Lloyd DP, Fiellin DA, Cutter CJ, Schottenfeld RS, Barry DT. Customized recommendations and reminder text messages for automated, computer-based treatment during methadone. Exp Clin Psychopharmacol. 2017 Dec;25(6):485-495. doi: 10.1037/pha0000149. PMID 29251978